CLINICAL TRIAL: NCT05923827
Title: Randomized Controlled Trial to Demonstrate the Efficacy of the Omnipod® 5 System When Compared to Multiple Daily Injections for Treatment of Type 1 Diabetes (RADIANT)
Brief Title: Omnipod® 5 With Libre 2 vs. MDI for Type 1 Diabetes in Children and Adults
Acronym: RADIANT
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Insulet Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RADIANT OP5-004
Record Dates: First submitted 2023-06-20; First posted 2023-06-28 (Actual); Last update posted 2024-10-26 (Actual); Status verified 2024-10

CONDITIONS: Diabetes Mellitus, Type 1
Keywords: T1D; Omnipod; Automated Insulin Delivery
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Intervention Group (Active Comparator): Omnipod 5 System with FreeStyle Libre 2 continuous glucose monitor
  Interventions: Device: Omnipod 5 System
- Control Group (No Intervention): Multiple daily injections of insulin with FreeStyle Libre 2 continuous glucose monitor

INTERVENTIONS:
Device: Omnipod 5 System — The Omnipod 5 system is a tubeless patch pump that receives glucose values and trend data from the glucose sensor every 5 minutes, automatically calculates insulin dose, and sends delivery commands to the Pod for the delivery of insulin.
  Arms: Intervention Group

SUMMARY:
This study is a randomized, controlled trial to evaluate the efficacy and safety of the Omnipod® 5 System with the FreeStyle Libre 2 continuous glucose monitor compared to Multiple Daily Injections (MDI) along with the FreeStyle Libre 2 continuous glucose monitor in children and adults with type 1.

DETAILED DESCRIPTION:
This is a prospective, randomized, parallel-group multicenter trial followed by an extension phase during which both groups use the Omnipod 5 system.

Participants will undergo a two-week standard therapy period utilizing the FreeStyle Libre 2 continuous glucose monitor (CGM) to collect baseline glycemic information.

Participants will then be randomized to the intervention or control groups (2:1).

Both groups will then participate in Period 1 for a total of 26-weeks after the completion of standard therapy period. During the first 13-weeks, participants randomized to the Control group will continue using MDI therapy with their Libre 2 CGM. Participants randomized to the Intervention group will onboard onto the Omnipod 5 System. At the conclusion of the 13-weeks, the Control group will onboard and use the Omnipod 5 System for an additional 13 weeks. Both groups will continue using the Omnipod 5 System for the remainder of the 26-weeks.

Participants in Belgium and France will be given the option to continue using the Omnipod 5 System for up to an additional 9-months.

ELIGIBILITY:
Inclusion Criteria:

1. Age at time of consent 4-70 years.
2. Clinical diagnosis of type 1 diabetes for at least 1 year prior to screening. Diagnosis is based on investigator's clinical judgement.
3. On MDI therapy (≥ 3 insulin injections per day and/or a basal/bolus regimen) for ≥ 3 months prior to screening. Have used insulin for at least 1 year prior to screening.
4. Have used the FreeStyle Libre 2 Sensor for ≥ 3 months with a daily average number of scans ≥ 4 and with sensor readings > 70% of time over the previous month prior to screening. Sensor usage is determined from the download summary report for 30 days preceding screening visit.
5. Must be willing to use the FreeStyle Libre 2 Sensor for the duration of the study.
6. HbA1c 7.5-11% (58-97mmol/mol) by point-of-care taken at screening visit
7. Deemed appropriate for pump therapy per investigator's assessment with respect to previous history of severe hypoglycemic and hyperglycemic events, other comorbidities, and capability of operating study devices and adhering to the protocol.
8. Willing to use and obtain U-100 insulin: either insulin aspart (Novolog, NovoRapid), or insulin lispro (Humalog, Admelog)) as the primary insulin treatment while using the Omnipod 5 System.
9. Participants or parent/guardian able to read and understand Dutch, English or French.
10. Willing to wear the system continuously throughout the study
11. Willing and able to sign the Informed Consent Form (ICF) and/or has a parent/guardian willing and able to sign the ICF. Assent will be obtained from pediatric and adolescent participants aged < 18 years per Country requirements.
12. Willing to limit vitamin C supplementation to 2000 mg or less per day.
13. Must be familiar with carbohydrate counting.

Exclusion Criteria:

1. Any medical condition, such as untreated malignancy, unstable cardiac disease, unstable or end-stage renal failure, eating disorders, or other conditions which in the opinion of the investigator, would put the participant at an unacceptable safety risk.
2. History of severe hypoglycemia in the past 6 months. Severe hypoglycemia is defined as an event that requires the assistance of another person due to altered consciousness, and requires another person to actively administer carbohydrate, glucagon, or other resuscitative actions.
3. History of diabetic ketoacidosis (DKA) in the past 6 months.
4. Blood disorder or dyscrasia within 3 months prior to screening, including use of hydroxyurea, which in the investigator's opinion could interfere with determination of HbA1c.
5. Using any form of pump therapy, including non-automated and automated insulin delivery (AID) systems, within 6 months prior to screening.
6. Currently on systemic steroids or intends to receive systemic steroid treatment in the next 6 months, including stable treatment for adrenal insufficiency. Inhaled, ophthalmic, topical, joint injection, and other locally applied steroids are allowed. If previously on oral steroids, last intake should be ≥14 days prior to screening visit.
7. Unable to tolerate adhesive tape or has any unresolved skin condition in the area of sensor or pump placement.
8. Use of non-insulin anti-hyperglycemic medication other than metformin, in the 12 weeks prior to the baseline visit and during the 6-month study. Participants taking metformin should remain on a steady dose during study participation.
9. Pregnant or lactating (lactating women are only excluded in France), or is a woman of childbearing potential and not on acceptable form of birth control (acceptable forms of contraception include abstinence, barrier methods such as condoms, hormonal contraceptives, intrauterine device, surgical sterilization such as tubal ligation or hysterectomy, or vasectomized partner).
10. Participation in another clinical study using an investigational drug or device within 30-days or 5 half-lives (whichever is longer) prior to screening, or intends to participate in any other drug or device study during this study period.
11. Unable to follow clinical protocol for the duration of the study or is otherwise deemed unacceptable to participate in the study per the investigator's clinical judgment.
12. Participant is an employee of Insulet, an Investigator or Investigator's study team, or immediate family member of any of the aforementioned.
13. Participants who have had a pancreas or pancreatic islet transplantation
14. Presence of unstable retinopathy or painful neuropathy, per Investigator's judgement.
15. Adult participants or parents/guardians with hearing and/or vision impairment that would interfere with recognition of all functions of the Omnipod 5 System, including alerts, alarms, and reminders.

Ages: 4 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2023-09-11 (Actual); Primary Completion 2024-08-02 (Actual); Study Completion 2025-08-08 (Estimated)

PRIMARY OUTCOMES:
Change in HbA1c | Comparing intervention group with control group during the 13-week study phase
  The change in HbA1c at 13 weeks from baseline between the Intervention and Control groups.

SECONDARY OUTCOMES:
Percentage of time in range 70-180 mg/dL | Comparing intervention group with control group during the 13-week study phase
  Glucose metric from study provided continuous glucose monitor (CGM)
Percentage of time <54 mg/dL (non-inferior) | Comparing intervention group with control group at the end of the 13-week study phase
  Glucose metric from CGM
Percentage of time >180 mg/dL | Comparing intervention group with control group at the end of the 13-week study phase
  Glucose metric from CGM
Percentage of time >300 mg/dL | Comparing intervention group with control group at the end of the 13-week study phase
  Glucose metric from CGM
Percentage of time <70 mg/dL (non-inferior) | Comparing intervention group with control group at the end of the 13-week study phase
  Glucose metric from CGM
Change from baseline in HbA1c for participants ≥18 years of age at baseline | Comparing intervention group with control group at the end of the 13-week study phase
  Glucose metric from study CGM
Change from baseline in HbA1c for participants <18 years of age at baseline | Comparing intervention group with control group at the end of the 13-week study phase
  Glucose metric from CGM
Percentage of time in range 70-180 mg/dL for participants ≥18 years of age at baseline | Comparing intervention group with control group at the end of the 13-week study phase
  Glucose metric from CGM
Percentage of time in range 70-180 mg/dL for participants <18 years of age at baseline | Comparing intervention group with control group at the end of the 13-week study phase
  Glucose metric from CGM
Change from baseline in HbA1c in participants with baseline HbA1c ≥8% | Comparing intervention group with control group at the end of the 13-week study phase
  Measured at baseline and 13 weeks in both intervention and control groups
Change from baseline in T1-DDS total score for participants ≥18 years of age at baseline | Comparing intervention group with control group at the end of the 13-week study phase
  A questionnaire that measures seven critical dimensions of distress (28-item scale with 6 choices that range from 1 (Not a Problem) to 6 (A Very Serious Problem)). The total score can range from 1 to 6, with a lower score indicating a better outcome.
Change from baseline in HCS total score for participants ≥18 years of age at baseline | Comparing intervention group with control group at the end of the 13-week study phase
  A questionnaire that examines the degree to which people with diabetes feel able, secure, and comfortable regarding their ability to stay safe from hypoglycemic-related problems (9-item scale with 4 choices that range from 1 (Not Confident At All) to 4 (Very Confident)). The total score can range from 1 to 4, with a higher score indicating a better outcome.
Change from baseline in PSQI Duration of Sleep subscale score in caregivers of participants <18 years of age at baseline | Comparing intervention group with control group at the end of the 13-week study phase
  Used to measure sleep disturbance and usual sleep habits
Change from baseline in PSQI Subjective Sleep Quality subscale score in caregivers of participants <18 years of age at baseline | Comparing intervention group with control group at the end of the 13-week study phase
  Used to measure sleep disturbance and usual sleep habits
Percentage of participants achieving HbA1c <7% | Comparing intervention group with control group at the end of the 13-week study phase
  Measured at 13 weeks in both intervention and control groups
Change from baseline in EQ-5D-3L index score | Comparing intervention group with control group at the end of the 13-week study phase
  Used to measure quality of life
Change from baseline in total daily insulin (TDI) (units/kg) for participants ≥18 years of age | Comparing intervention group with control group at the end of the 13-week study phase
  Measure of insulin requirements measured at 13 weeks in both intervention and control groups
Percentage of time <70 mg/dL | Comparing intervention group with control group at the end of the 13-week study phase
  Glucose metric from CGM
Percentage of time <54 mg/dL | Comparing intervention group with control group at the end of the 13-week study phase
  Glucose metric from CGM

CONTACTS AND LOCATIONS:
Overall Officials: Emma Wilmot, MD, Principal Investigator — University Hospitals of Derby & Burton NHS Foundation Trust
Locations (19):
- Belgium (2):
  - Cliniques Universitaires Saint-Luc, Brussels
  - Universitaire Ziekenhuizen Leuven, Leuven
- France (12):
  - Centre Hospitalier Universitaire Côte de Nacre, Caen
  - CHU Grenoble Aples, Grenoble
  - Hospices Civils de Lyon, Lyon
  - Hôpitaux Universitaires de Marseille Timone, Marseille
  - CHU de Nancy, Nancy
  - Hôpitaux Pédiatriques de Nice CHU-Lenval,, Nice
  - Centre Hospitalier Universitaire Carémeau de Nîmes, Nîmes
  - Hôpital Necker, Paris
  - Robert-Debré AP-HP Hospital, Paris
  - Centre Hospitalier Universitaire de Reims, Reims
  - CHU Rennes, Rennes
  - CHU Toulouse, Toulouse
- United Kingdom (5):
  - University Hospitals of Derby & Burton, Derby
  - University Hospitals of Leicester NHS Trust, Leicester
  - Manchester University NHS Foundation Trust, Manchester
  - Mersey and West Lancashire NHS Teaching Hospitals Trust, Ormskirk
  - Oxford Health NHS Foundation Trust, Oxford

IPD SHARING:
Plan to Share IPD: No